CLINICAL TRIAL: NCT00827203
Title: A Phase 1 Multi-Dose Dose-Escalation Study of Elesclomol Sodium, Administered Once Weekly to Subjects With Solid Tumors
Brief Title: A Safety Study to Determine the Maximum Tolerated Dose of Elesclomol Sodium in Patients With Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: David Hynds, Clinical Trials Manager, Synta Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4783-11
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Metastatic Solid Tumors
Keywords: cancer; metastatic; Elesclomol Sodium; tumor; Advanced solid tumors that are metastatic and unresectable
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Experimental)
  Interventions: Drug: Elesclomol Sodium

INTERVENTIONS:
Drug: Elesclomol Sodium — Chemotherapy agent

SUMMARY:
The aim of this study is to determine the safety and tolerability of elesclomol sodium at escalating doses (ultimately identifying the maximum tolerated dose). This study will also characterize the pharmacokinetics of elesclomol and evaluate its anti-tumor activity in advanced solid tumors that are metastatic and unresectable.

ELIGIBILITY:
Inclusion Criteria

* Males and females at least 18 years of age
* Histologically- or cytologically- confirmed solid tumor (except melanoma) that is metastatic or unresectable
* Advanced or metastatic cancer for which no standard therapy exists or that has progressed despite standard therapy
* Acceptable organ and marrow function during the Screening Period as defined by the protocol.
* Reliable venous access suitable for weekly study drug infusions
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria

* Pregnant or breast-feeding women
* Have had chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Primary brain tumors or active brain metastases
* Treatment with chronic immunosuppressants
* Significant cardiovascular disease, severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of elesclomol sodium administered once weekly to subjects with solid tumors | Jan 2011
To determine the pharmacokinetics of elesclomol in this population when administered once weekly as a 1-hour intravenous infusion | Jan 2011

SECONDARY OUTCOMES:
To inform dose selection for future study using a once-a-week schedule | Jan 2011
To evaluate anti-tumor activity in advanced solid tumors that are metastatic and unresectable | Jan 2011
To assess the effect of elesclomol sodium on the development of peripheral neuropathy by rating sensory symptoms, strength, tendon reflexes, and vibratory sense | Jan 2011

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Maryland
  - University of Texas Health Science Center, Cancer Therapy & Research Center, Institute for Drug Development, San Antonio, Texas
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin